CLINICAL TRIAL: NCT00005919
Title: Etiology of Pigment Dispersion Syndrome (PDS)
Brief Title: Cause of Pigment Dispersion Syndrome
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000155; 00-EI-0155
Record Dates: First submitted 2000-06-17; First posted 2000-06-19 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-08

CONDITIONS: Glaucoma; Healthy; Pigment Dispersion Syndrome
Keywords: Pigment Dispersion; Ocular Hypertension; Glaucoma; Pupil Reaction; Natural History; Pigment Dispersion Syndrome; Gene Mutation
MeSH Terms: conditions — Glaucoma; Glaucoma-Related Pigment Dispersion Syndrome; Ocular Hypertension

SUMMARY:
The purpose of this study is to learn how pigment is released from the iris (the colored part of the eye) in patients with pigment dispersion syndrome. It will do this by examining the response of the pupil (the central opening of the iris) to a flash of light to determine what is happening in the iris to cause release of the pigment.

In pigment dispersion syndrome, pigment released from the iris is deposited in other parts of the eye, including the trabecular meshwork-a filter-like tissue in the front of the eye. Aqueous fluid (fluid continuously produced by the eye) normally flows out of the eye through the trabecular meshwork. In some patients, the pigment deposits may block tiny holes in the meshwork, preventing the fluid from flowing out. This can cause an increase in eye pressure that may lead to glaucoma and some loss of vision. Understanding how pigment is released from the iris may help predict the course of pigment dispersion syndrome and identify which patients will likely develop increased eye pressure.

Patients with pigment dispersion syndrome and normal volunteers may be eligible for this study. All participants will have the following procedures, which will be completed in two clinic visits:

First visit

1. Examination of the front of the eyes, including the cornea, iris and lens.
2. Vision testing and measurements of visual field and eye pressure.
3. Examination of the trabecular meshwork. For this test, a contact lens is placed on the eye after the eye has been numbed with anesthetic drops.

Second visit

1. Refraction (dilation of the pupils with drops) and examination of the back of the eyes, including the optic nerve.
2. Reaction of the pupils to low-level infrared light (pupillography). During this 15-minute test, the patient or volunteer wears a lightweight headband with two small cameras mounted on it. The cameras-one which views the eye and the other the subject's field of view-record pupil dilation and position.

The test results in patients with pigment dispersion syndrome will be compared with those in normal volunteers. Patients will be followed every 6 months (or more often, if medically indicated) during the 3-year study to determine changes in eye pressure or visual field. Volunteers will be asked to return about once a year for 3 years for repeat pupillography.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a comprehensive ophthalmologic evaluation and comparison of two types of patients and to compare them to normal controls. The two types of patients are those with pigment dispersion (PDS) with normal intraocular pressure (IOP) and those with PDS and elevated IOP. The hypothesis to be tested is that a developmental abnormality of the iris pigment epithelium (IPE) and the dilator muscle is the fundamental defect responsible for the pigment dispersion. This defect may involve other structures of the eye such as the ciliary and retinal pigment epithelium. The results of pupillography in PDS with or without elevated IOP and asymmetric PDS (one eye versus fellow eye) will be the outcome parameters.

ELIGIBILITY:
INCLUSION CRITERIA:

All patients entering the study must have black pigment deposition on the trabecular meshwork at the site of Schlemm's canal equal to or greater than 2-plus on the goniophotographic scale of 1 to 5 plus.

Although this condition is rare amongst African-Americans, every effort will be made to recruit such individuals.

EXCLUSION CRITERIA:

Patients with exfoliation syndrome, uveitis, trauma, pigment dispersion with posterior chamber intra-ocular lens, pigmented tumors, primary open-angle glaucoma, other conditions with associated pigment dispersion such as acute angle-closure glaucoma, ocular hemorrhage, Horner's syndrome.

In addition, normal volunteers will be recruited as controls. They will be free of any eye disease and be matched for age, sex and degree of myopia.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 2000-06; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ferris FL 3rd, Sperduto RD. Standardized illumination for visual acuity testing in clinical research. Am J Ophthalmol. 1982 Jul;94(1):97-8. doi: 10.1016/0002-9394(82)90198-2. No abstract available. PMID 7091290
- [Background] Ferris FL 3rd, Kassoff A, Bresnick GH, Bailey I. New visual acuity charts for clinical research. Am J Ophthalmol. 1982 Jul;94(1):91-6. PMID 7091289